CLINICAL TRIAL: NCT01280760
Title: Impact of Neurally Adjusted Ventilator Assist (NAVA) Mode on Patient Ventilator Asynchrony Using Non-invasive Ventilation (NAVA-NIV)
Acronym: NAVA-NIV
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Matthieu SCHMIDT, Dr, Pierre and Marie Curie University
Other Study IDs: UPMC
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Weaning Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non invasive ventilation: Non-invasive ventilation after invasive mechanical ventilation weaning
  Interventions: Other: Device: Neurally Adjusted Ventilatory Assistance

INTERVENTIONS:
Other: Device: Neurally Adjusted Ventilatory Assistance — Device: Neurally Adjusted Ventilatory Assistance
  In ICU following extubation NIV was performed as follows:
  facial mask with PSV/NIV mode to define settings for NAVA ventilation facial use with NAVA/NIV mode

SUMMARY:
Non-invasive ventilation (NIV) has been proposed to reduce the incidence of ventilatory dysfunction following mechanical ventilation weaning. However, the nasogastric tube reduces the airtightness of the facial mask used to perform non-invasive ventilation and induces air leaks. The presence of leaks at the patient-mask interface can increase the risk of patient-ventilator asynchrony, which in turn leads to increase patient discomfort. Neurally adjusted ventilatory assist (NAVA)could contribute to decreasing asynchrony. Its principle is to record the diaphragmatic electrical activity and to control the ventilator. The investigators hypothesized driving the ventilator based on a neural signal (diaphragm electrical activity) would reduce patient-ventilator asynchronies in NIV

ELIGIBILITY:
Inclusion Criteria:

Patients with increased risk of post-extubation ventilatory dysfunction following invasive mechanical ventilation weaning.

Exclusion Criteria:

* Contra-indication to non-invasive ventilation
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NIV required on post extubation period
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Triggering delay | Every inspiration, for 10 minutes
  Duration between the onset of neural inspiration and the onset of insufflation

SECONDARY OUTCOMES:
Cycling off delay | Every inspiration, for 10 minutes
  Delay between the end of neural inspiration and the end of insufflation

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Pitié Salpétrière, Department of intensive care and pneumology, Paris, France

REFERENCES:
- [Derived] Schmidt M, Dres M, Raux M, Deslandes-Boutmy E, Kindler F, Mayaux J, Similowski T, Demoule A. Neurally adjusted ventilatory assist improves patient-ventilator interaction during postextubation prophylactic noninvasive ventilation. Crit Care Med. 2012 Jun;40(6):1738-44. doi: 10.1097/CCM.0b013e3182451f77. PMID 22610179